CLINICAL TRIAL: NCT00481221
Title: Detection of β Thalassemia Carriers by Red Cell Parameters Obtained From the H2 Automatic Counter. A Clinical Retrospective Study.
Brief Title: Detection of β Thalassemia Carriers by Red Cell Parameters Obtained From the H2 Automatic Counter
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Hematology Unit and Pediatric Dpt B, HaEmek Medical Center, Israel
Other Study IDs: 5210906.EMC
Record Dates: First submitted 2007-05-31; First posted 2007-06-01 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Thalassemia; Iron Deficiency
Keywords: Thalassemia; Iron Deficiency; Carrier screening
MeSH Terms: conditions — Thalassemia; Iron Deficiencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Screened pregnant women
  Interventions: Procedure: Observation of results from laboratory tests

INTERVENTIONS:
Procedure: Observation of results from laboratory tests — Laboratory data summary only

SUMMARY:
β thalassemia is an autosomal recessive hemoglobinopathy and considered as the most widespread genetic mutation. According to the World Health Organization (WHO) between 1.5-7% of the world population are carriers for this disease, and every year 60,000-400,000 birth of new patients are reported. In Israel, the incidence of carriers for β thalassemia is around 20% among the Jewish from Kurdish origin and around 5-10% among the Arab population.

β thalassemia is a severe disease which requires many resources, both medical and financial. The disease is expressed by chronic hemolytic anemia which requires regular blood transfusions every 3 weeks. As a result of the blood transfusions and the iron absorption by the digestive tract, those patients suffer from severe hemosiderosis which is the main mortality cause in the disease, mainly in the second decade for life. Daily treatment with iron chelator is required. Moreover, despite the actual treatment, the quality of life of those patients is still low.

Therefore the implementation of a prevention program which includes finding an effective and inexpensive way for identifying the β thalassemia carriers is a humanitary and publicly important goal.

In β thalassemia carriers, laboratory tests will show hypochromic microcytic anemia. Those findings are similar in iron deficiency anemia, but the RBC number and the RDW are normal in thalassemia carriers.

Few researchers tried in the past to determine cutoff point for diagnosis of β thalassemia carriers by different formulas.

We used the algorithm SVM (support vector machine) to find a reliable formula that can separate patients with Iron deficiency anemia/ healthy from patients with β thalassemia minor (carriers). This formula can be inserted to any automatic blood counter and search for suspected carriers without deliberately intention and without any further blood test.

ELIGIBILITY:
Inclusion Criteria:

* Blood count and Hgb electrophoresis analysis received from pregnant women send for screening for thalassemia.

Exclusion Criteria:

* Age below 17 yrs and older than 50 yrs.
* Sever anemia with hgb level below 8 gr/dl.

Ages: 17 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All pregant women attending to the Mother's and Child stations in northern Israel
Sampling Method: Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2007-03; Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of β Thalassemia Carriers by Red Cell Parameters | One year
  Detection of β Thalassemia Carriers by Red Cell Parameters Obtained From the Automatic blood count counter using mathematics formula

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Koren, MD, Study Director — Pediatric Hematology Unit, Ha'Emek Medical Center; Idit Koren, Medical Student, Principal Investigator — Pediatric Hematology Unit - Ha'Emek Medical Center; Carina Levin, MD, Study Chair — Pediatric Dpt B - Ha'Emek Medical Center; Luci Zalman, PhD, Study Chair — Hematology Laboratory - HaEmek Medical Center
Locations (1):
- Pediatric Hematology Unit - HaEmek Medical Center, Afula, Israel